CLINICAL TRIAL: NCT03976466
Title: Application of Antibiotic Loaded Calcium Sulfate as Prophylaxis for Patients With Non Modifiable Risk Factors for Periprosthetic Joint Infections
Brief Title: Prophylaxis of Periprosthetic Joint Infections With Calcium Sulfate Beads in Patients With Non-modifiable Risk Factors.
Acronym: Stimulan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Regional Tlalnepantla (Other Government)
Responsible Party: Principal Investigator, Julio Carlos Velez de Lachica, Md. High Specialty Associate Professor of the Joint Surgery Course., Hospital Regional Tlalnepantla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Infection
Keywords: Periprosthetic Joint Infection; Prophylaxis; Joint Replacement; Calcium Sulfate Beads
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Study participants are randomly assigned to one of two groups: the experimental group receiving the Calcium sulfate beds with antibiotics and a comparison group (control) which receives a conventional prophylactic therapy.
Who Masked: Participant
Masking Description: No participant will know during the study in which group will be assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium sulfate Group (Experimental): Group of members that will be submitted to prophylaxis with medicated calcium sulfate beads for hip or knee joint replacement
  Interventions: Device: Antibiotic local prophylaxis with medicated calcium sulfate beads
- Control Group (Active Comparator): Group of members that will be submitted to classic prophylaxis for hip or knee joint replacement
  Interventions: Procedure: Classical parenteral antibiotic prophylaxis

INTERVENTIONS:
Device: Antibiotic local prophylaxis with medicated calcium sulfate beads — Antibiotic prophylaxis in patients with non-modifiable risk factors for periprosthetic joint infection
  Other Names: Hip or Knee Joint Replacement
  Arms: Calcium sulfate Group
Procedure: Classical parenteral antibiotic prophylaxis — Antibiotic prophylaxis in patients with non-modifiable risk factors for periprosthetic joint infection
  Other Names: Hip pr Knee Joint Replacement
  Arms: Control Group

SUMMARY:
To demonstrate the prophylactic effect of calcium sulfate beads loaded with antibiotic in patients with non-modifiable risk factors that will undergo a hip or knee joint replacement, comparing with a control group.

To know the economic cost generated in antibiotic prophylaxis with calcium sulfate beads in patients undergoing hip or knee joint replacement with non-modifiable risk factors.

DETAILED DESCRIPTION:
Since joint replacement procedures have been successful in recent decades, every year the number of implanted prostheses is increasing, however, at the same time, orthopaedic surgeons also find complications inherent to this surgery, where peri-prosthetic infection results to be the most devastating. In order to find a solution to this terrible complication, prophylactic and therapeutic measures have been implemented, emerging techniques where the application of local antibiotics in the surgical site has turned out to be a promising concept. It has been shown that the non-modifiable risk factors of patients undergoing joint replacement surgery increase the risk of infection rate. Therefore, the identification of risk factors, decolonization and the prophylactic administration of antibiotics allow an effective reduction of periprosthetic infection. In order to reduce and, as far as posible, avoid periprosthetic infections in participants undergo knee or hip joint replacement with non-modifiable risk factors, the prophylactic use of calcium sulphate loaded with antibiotic for local application is proposed.

ELIGIBILITY:
Inclusion Criteria:

* patients with fracture or osteoarthrosis of the hip or knee that require treatment by joint replacement.
* patients who have any of the Non-Modifiable Risk Factors prior to surgery or during transoperative period.
* Patients entitled to the ISSEMyM (Instituto de Seguridad Social del Estado de Mexico y Municipios)

Exclusion Criteria:

* Patients that lose their validity of institutional rights and do not follow up
* Patients who die during the study due to other causes not related to the orthopedic procedure.
* Patients who do not have any of the risk factors for periprosthetic infection
* Patients allergic to vancomycin or ceftriaxone.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HOSPITAL REGIONAL TLALNEPANTLA ISSEMyM, Tlalnepantla, Mexico

REFERENCES:
- [Background] Ong KL, Kurtz SM, Lau E, Bozic KJ, Berry DJ, Parvizi J. Prosthetic joint infection risk after total hip arthroplasty in the Medicare population. J Arthroplasty. 2009 Sep;24(6 Suppl):105-9. doi: 10.1016/j.arth.2009.04.027. Epub 2009 Jun 2. PMID 19493644
- [Background] Pulido L, Ghanem E, Joshi A, Purtill JJ, Parvizi J. Periprosthetic joint infection: the incidence, timing, and predisposing factors. Clin Orthop Relat Res. 2008 Jul;466(7):1710-5. doi: 10.1007/s11999-008-0209-4. Epub 2008 Apr 18. PMID 18421542
- [Background] Wahl P, Guidi M, Benninger E, Ronn K, Gautier E, Buclin T, Magnin JL, Livio F. The levels of vancomycin in the blood and the wound after the local treatment of bone and soft-tissue infection with antibiotic-loaded calcium sulphate as carrier material. Bone Joint J. 2017 Nov;99-B(11):1537-1544. doi: 10.1302/0301-620X.99B11.BJJ-2016-0298.R3. PMID 29092996
- [Background] Wahl P, Livio F, Jacobi M, Gautier E, Buclin T. Systemic exposure to tobramycin after local antibiotic treatment with calcium sulphate as carrier material. Arch Orthop Trauma Surg. 2011 May;131(5):657-62. doi: 10.1007/s00402-010-1192-2. Epub 2010 Oct 12. PMID 20938669
- [Background] Reed EE, Johnston J, Severing J, Stevenson KB, Deutscher M. Nephrotoxicity Risk Factors and Intravenous Vancomycin Dosing in the Immediate Postoperative Period Following Antibiotic-Impregnated Cement Spacer Placement. Ann Pharmacother. 2014 Aug;48(8):962-969. doi: 10.1177/1060028014535360. Epub 2014 May 13. PMID 24823910
- [Background] Horii C, Yamazaki T, Oka H, Azuma S, Ogihara S, Okazaki R, Kawamura N, Takano Y, Morii J, Takeshita Y, Maruyama T, Yamakawa K, Murakami M, Oshima Y, Tanaka S. Does intrawound vancomycin powder reduce surgical site infection after posterior instrumented spinal surgery? A propensity score-matched analysis. Spine J. 2018 Dec;18(12):2205-2212. doi: 10.1016/j.spinee.2018.04.015. Epub 2018 Apr 26. PMID 29705336
- [Background] Sweet FA, Roh M, Sliva C. Intrawound application of vancomycin for prophylaxis in instrumented thoracolumbar fusions: efficacy, drug levels, and patient outcomes. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2084-8. doi: 10.1097/BRS.0b013e3181ff2cb1. PMID 21304438
- [Background] Zebala LP, Chuntarapas T, Kelly MP, Talcott M, Greco S, Riew KD. Intrawound vancomycin powder eradicates surgical wound contamination: an in vivo rabbit study. J Bone Joint Surg Am. 2014 Jan 1;96(1):46-51. doi: 10.2106/JBJS.L.01257. PMID 24382724
- [Background] Whiteside LA, Peppers M, Nayfeh TA, Roy ME. Methicillin-resistant Staphylococcus aureus in TKA treated with revision and direct intra-articular antibiotic infusion. Clin Orthop Relat Res. 2011 Jan;469(1):26-33. doi: 10.1007/s11999-010-1313-9. PMID 20390472
- [Background] Buchholz HW, Engelbrecht H. [Depot effects of various antibiotics mixed with Palacos resins]. Chirurg. 1970 Nov;41(11):511-5. No abstract available. German. PMID 5487941
- [Background] Bennett-Guerrero E, Pappas TN, Koltun WA, Fleshman JW, Lin M, Garg J, Mark DB, Marcet JE, Remzi FH, George VV, Newland K, Corey GR; SWIPE 2 Trial Group. Gentamicin-collagen sponge for infection prophylaxis in colorectal surgery. N Engl J Med. 2010 Sep 9;363(11):1038-49. doi: 10.1056/NEJMoa1000837. Epub 2010 Aug 4. PMID 20825316
- [Background] Birgand G, Radu C, Alkhoder S, Al Attar N, Raffoul R, Dilly MP, Nataf P, Lucet JC. Does a gentamicin-impregnated collagen sponge reduce sternal wound infections in high-risk cardiac surgery patients? Interact Cardiovasc Thorac Surg. 2013 Feb;16(2):134-41. doi: 10.1093/icvts/ivs449. Epub 2012 Oct 31. PMID 23115102
- [Background] KOVACEVIC B. [Problem of hematogenous osteomyelitis]. Langenbecks Arch Klin Chir Ver Dtsch Z Chir. 1953;276:432-43. No abstract available. Undetermined Language. PMID 13143827
- [Background] Fischer G, Seidler W. [Results in the treatment of osteomyelitic bone cavities using antibiotic gypsum medullary plombage]. Dtsch Gesundheitsw. 1971 Nov 4;26(45):2105-7. No abstract available. German. PMID 5145654
- [Background] Mackey D, Varlet A, Debeaumont D. Antibiotic loaded plaster of Paris pellets: an in vitro study of a possible method of local antibiotic therapy in bone infection. Clin Orthop Relat Res. 1982 Jul;(167):263-8. PMID 7094471
- [Background] Varlet A, Dauchy P. [Plaster of Paris pellets containing antibiotics in the treatment of bone infection. New combinations of plaster with antibiotics]. Rev Chir Orthop Reparatrice Appar Mot. 1983;69(3):239-44. French. PMID 6224275
- [Background] Dahners LE, Funderburk CH. Gentamicin-loaded plaster of Paris as a treatment of experimental osteomyelitis in rabbits. Clin Orthop Relat Res. 1987 Jun;(219):278-82. PMID 3581579
- [Background] Evrard J, Kerri O, Martini M, Conort O. [Treatment of bone infection by plaster of Paris pellets impregnated with antibiotics]. Pathol Biol (Paris). 1990 Jun;38(5 ( Pt 2)):543-7. French. PMID 2385452
- [Background] Mousset B, Benoit MA, Bouillet R, Gillard J. [Plaster of Paris: a carrier for antibiotics in the treatment of bone infections]. Acta Orthop Belg. 1993;59(3):239-48. French. PMID 8237338
- [Background] Sulo I. [Gentamycin impregnated plaster beads in the treatment of bone infection]. Rev Chir Orthop Reparatrice Appar Mot. 1993;79(4):299-305. French. PMID 8159845
- [Background] Gitelis S, Brebach GT. The treatment of chronic osteomyelitis with a biodegradable antibiotic-impregnated implant. J Orthop Surg (Hong Kong). 2002 Jun;10(1):53-60. doi: 10.1177/230949900201000110. PMID 12401922
- [Background] Meza-Lopez LR, Cigarroa-Lopez JA, Hernandez-Meneses S, Castan-Flores DA, Mendoza-Zavala GH, Barragan-Zamora JA, Carrillo-Munoz A, Munguia-Canales DA. [Dissolvable and extended release antibiotic beads in mediastinoscopic management of mediastinitis after heart transplantation]. Arch Cardiol Mex. 2017 Apr-Jun;87(2):182-186. doi: 10.1016/j.acmx.2017.01.006. Epub 2017 Mar 2. No abstract available. Spanish. PMID 28259393
- [Background] Aiken SS, Cooper JJ, Florance H, Robinson MT, Michell S. Local release of antibiotics for surgical site infection management using high-purity calcium sulfate: an in vitro elution study. Surg Infect (Larchmt). 2015 Feb;16(1):54-61. doi: 10.1089/sur.2013.162. Epub 2014 Aug 22. PMID 25148101
- [Background] Howlin RP, Brayford MJ, Webb JS, Cooper JJ, Aiken SS, Stoodley P. Antibiotic-loaded synthetic calcium sulfate beads for prevention of bacterial colonization and biofilm formation in periprosthetic infections. Antimicrob Agents Chemother. 2015 Jan;59(1):111-20. doi: 10.1128/AAC.03676-14. Epub 2014 Oct 13. PMID 25313221
- [Background] Howlin RP, Winnard C, Angus EM, Frapwell CJ, Webb JS, Cooper JJ, Aiken SS, Bishop JY, Stoodley P. Prevention of Propionibacterium acnes biofilm formation in prosthetic infections in vitro. J Shoulder Elbow Surg. 2017 Apr;26(4):553-563. doi: 10.1016/j.jse.2016.09.042. Epub 2016 Dec 15. PMID 27989720
- [Background] Howlin RP, Winnard C, Frapwell CJ, Webb JS, Cooper JJ, Aiken SS, Stoodley P. Biofilm prevention of gram-negative bacterial pathogens involved in periprosthetic infection by antibiotic-loaded calcium sulfate beads in vitro. Biomed Mater. 2016 Dec 2;12(1):015002. doi: 10.1088/1748-605X/12/1/015002. PMID 27910828
- [Background] Kallala R, Harris WE, Ibrahim M, Dipane M, McPherson E. Use of Stimulan absorbable calcium sulphate beads in revision lower limb arthroplasty: Safety profile and complication rates. Bone Joint Res. 2018 Nov 3;7(10):570-579. doi: 10.1302/2046-3758.710.BJR-2017-0319.R1. eCollection 2018 Oct. PMID 30464837
- [Background] Lum ZC, Pereira GC. Local bio-absorbable antibiotic delivery in calcium sulfate beads in hip and knee arthroplasty. J Orthop. 2018 May 7;15(2):676-678. doi: 10.1016/j.jor.2018.05.001. eCollection 2018 Jun. PMID 29881219
- [Background] Kurtz SM, Lau E, Watson H, Schmier JK, Parvizi J. Economic burden of periprosthetic joint infection in the United States. J Arthroplasty. 2012 Sep;27(8 Suppl):61-5.e1. doi: 10.1016/j.arth.2012.02.022. Epub 2012 May 2. PMID 22554729
- [Background] Parvizi J, Pawasarat IM, Azzam KA, Joshi A, Hansen EN, Bozic KJ. Periprosthetic joint infection: the economic impact of methicillin-resistant infections. J Arthroplasty. 2010 Sep;25(6 Suppl):103-7. doi: 10.1016/j.arth.2010.04.011. Epub 2010 May 31. PMID 20570103
- [Background] Parvizi J, Azzam K, Ghanem E, Austin MS, Rothman RH. Periprosthetic infection due to resistant staphylococci: serious problems on the horizon. Clin Orthop Relat Res. 2009 Jul;467(7):1732-9. doi: 10.1007/s11999-009-0857-z. Epub 2009 May 1. PMID 19408061
- [Background] Kurtz SM, Lau E, Schmier J, Ong KL, Zhao K, Parvizi J. Infection burden for hip and knee arthroplasty in the United States. J Arthroplasty. 2008 Oct;23(7):984-91. doi: 10.1016/j.arth.2007.10.017. Epub 2008 Apr 10. PMID 18534466
- [Background] Almeida Herrero F, Lopez Lozano R, Silvestre Munoz A. [Descriptive analysis of C-Reactive values after uncomplicated total hip and knee arthroplasty]. Acta Ortop Mex. 2008 Mar-Apr;22(2):80-4. Spanish. PMID 18669307
- [Background] Bilgen O, Atici T, Durak K, Karaeminogullari, Bilgen MS. C-reactive protein values and erythrocyte sedimentation rates after total hip and total knee arthroplasty. J Int Med Res. 2001 Jan-Feb;29(1):7-12. doi: 10.1177/147323000102900102. PMID 11277348
- [Background] Greidanus NV, Masri BA, Garbuz DS, Wilson SD, McAlinden MG, Xu M, Duncan CP. Use of erythrocyte sedimentation rate and C-reactive protein level to diagnose infection before revision total knee arthroplasty. A prospective evaluation. J Bone Joint Surg Am. 2007 Jul;89(7):1409-16. doi: 10.2106/JBJS.D.02602. PMID 17606776
- [Background] Hashmi FR, Barlas K, Mann CF, Howell FR. Staged bilateral hip or knee arthroplasties. J Orthop Surg (Hong Kong). 2007 Aug;15(2):159-62. doi: 10.1177/230949900701500206. PMID 17709852
- [Background] Larsson S, Thelander U, Friberg S. C-reactive protein (CRP) levels after elective orthopedic surgery. Clin Orthop Relat Res. 1992 Feb;(275):237-42. PMID 1735220
- [Background] Nazem K, Motififard M, Yousefian M. Variations in ESR and CRP in total knee arthroplasty and total hip arthroplasty in Iranian patients from 2009 to 2011. Adv Biomed Res. 2016 Aug 30;5:148. doi: 10.4103/2277-9175.187403. eCollection 2016. PMID 27656617
- [Background] Park KK, Kim TK, Chang CB, Yoon SW, Park KU. Normative Temporal Values of CRP and ESR in Unilateral and Staged Bilateral TKA. Clin Orthop Relat Res. 2008 Jan;466(1):179-88. doi: 10.1007/s11999-007-0001-x. Epub 2008 Jan 3. PMID 18196391
- [Background] Parvizi J, Ghanem E, Sharkey P, Aggarwal A, Burnett RS, Barrack RL. Diagnosis of infected total knee: findings of a multicenter database. Clin Orthop Relat Res. 2008 Nov;466(11):2628-33. doi: 10.1007/s11999-008-0471-5. Epub 2008 Sep 10. PMID 18781372
- [Background] White J, Kelly M, Dunsmuir R. C-reactive protein level after total hip and total knee replacement. J Bone Joint Surg Br. 1998 Sep;80(5):909-11. doi: 10.1302/0301-620x.80b5.8708. PMID 9768908
- [Background] Yi PH, Cross MB, Moric M, Sporer SM, Berger RA, Della Valle CJ. The 2013 Frank Stinchfield Award: Diagnosis of infection in the early postoperative period after total hip arthroplasty. Clin Orthop Relat Res. 2014 Feb;472(2):424-9. doi: 10.1007/s11999-013-3089-1. PMID 23884798
- [Background] Zimmerli W. Clinical presentation and treatment of orthopaedic implant-associated infection. J Intern Med. 2014 Aug;276(2):111-9. doi: 10.1111/joim.12233. PMID 24605880
- [Background] Arnold WV, Shirtliff ME, Stoodley P. Bacterial biofilms and periprosthetic infections. J Bone Joint Surg Am. 2013 Dec 18;95(24):2223-9. doi: 10.2106/JBJS.2223. No abstract available. PMID 24498639
- [Background] McConoughey SJ, Howlin R, Granger JF, Manring MM, Calhoun JH, Shirtliff M, Kathju S, Stoodley P. Biofilms in periprosthetic orthopedic infections. Future Microbiol. 2014;9(8):987-1007. doi: 10.2217/fmb.14.64. PMID 25302955
- [Background] Arciola CR, Campoccia D, Montanaro L. Implant infections: adhesion, biofilm formation and immune evasion. Nat Rev Microbiol. 2018 Jul;16(7):397-409. doi: 10.1038/s41579-018-0019-y. PMID 29720707
- [Background] Klemm K. [Gentamicin-PMMA-beads in treating bone and soft tissue infections (author's transl)]. Zentralbl Chir. 1979;104(14):934-42. German. PMID 494865
- [Background] Nelson CL, Jones RB, Wingert NC, Foltzer M, Bowen TR. Sonication of antibiotic spacers predicts failure during two-stage revision for prosthetic knee and hip infections. Clin Orthop Relat Res. 2014 Jul;472(7):2208-14. doi: 10.1007/s11999-014-3571-4. PMID 24658903
- [Background] Neut D, van de Belt H, Stokroos I, van Horn JR, van der Mei HC, Busscher HJ. Biomaterial-associated infection of gentamicin-loaded PMMA beads in orthopaedic revision surgery. J Antimicrob Chemother. 2001 Jun;47(6):885-91. doi: 10.1093/jac/47.6.885. PMID 11389124
- [Background] Tunney MM, Ramage G, Patrick S, Nixon JR, Murphy PG, Gorman SP. Antimicrobial susceptibility of bacteria isolated from orthopedic implants following revision hip surgery. Antimicrob Agents Chemother. 1998 Nov;42(11):3002-5. doi: 10.1128/AAC.42.11.3002. PMID 9797241
- [Background] Chang CC, Merritt K. Microbial adherence on poly(methyl methacrylate) (PMMA) surfaces. J Biomed Mater Res. 1992 Feb;26(2):197-207. doi: 10.1002/jbm.820260206. PMID 1569113
- [Background] Saginur R, Stdenis M, Ferris W, Aaron SD, Chan F, Lee C, Ramotar K. Multiple combination bactericidal testing of staphylococcal biofilms from implant-associated infections. Antimicrob Agents Chemother. 2006 Jan;50(1):55-61. doi: 10.1128/AAC.50.1.55-61.2006. PMID 16377667
- [Background] van de Belt H, Neut D, Schenk W, van Horn JR, van der Mei HC, Busscher HJ. Infection of orthopedic implants and the use of antibiotic-loaded bone cements. A review. Acta Orthop Scand. 2001 Dec;72(6):557-71. doi: 10.1080/000164701317268978. PMID 11817870
- [Background] Winkler H. Treatment of chronic orthopaedic infection. EFORT Open Rev. 2017 May 11;2(5):110-116. doi: 10.1302/2058-5241.2.160063. eCollection 2017 May. PMID 28630748
- [Background] Zhu Y, Zhang F, Chen W, Liu S, Zhang Q, Zhang Y. Risk factors for periprosthetic joint infection after total joint arthroplasty: a systematic review and meta-analysis. J Hosp Infect. 2015 Feb;89(2):82-9. doi: 10.1016/j.jhin.2014.10.008. Epub 2014 Dec 4. PMID 25575769
- [Background] Cordero-Ampuero J, de Dios M. What are the risk factors for infection in hemiarthroplasties and total hip arthroplasties? Clin Orthop Relat Res. 2010 Dec;468(12):3268-77. doi: 10.1007/s11999-010-1411-8. PMID 20544319
- [Background] Namba RS, Inacio MC, Paxton EW. Risk factors associated with deep surgical site infections after primary total knee arthroplasty: an analysis of 56,216 knees. J Bone Joint Surg Am. 2013 May 1;95(9):775-82. doi: 10.2106/JBJS.L.00211. PMID 23636183
- [Background] Neut D, van de Belt H, van Horn JR, van der Mei HC, Busscher HJ. Residual gentamicin-release from antibiotic-loaded polymethylmethacrylate beads after 5 years of implantation. Biomaterials. 2003 May;24(10):1829-31. doi: 10.1016/s0142-9612(02)00614-2. PMID 12593965
- [Background] Wilson KJ, Cierny G, Adams KR, Mader JT. Comparative evaluation of the diffusion of tobramycin and cefotaxime out of antibiotic-impregnated polymethylmethacrylate beads. J Orthop Res. 1988;6(2):279-86. doi: 10.1002/jor.1100060216. PMID 3278081
- [Background] Ribeiro M, Monteiro FJ, Ferraz MP. Infection of orthopedic implants with emphasis on bacterial adhesion process and techniques used in studying bacterial-material interactions. Biomatter. 2012 Oct-Dec;2(4):176-94. doi: 10.4161/biom.22905. PMID 23507884
- [Background] Rimondini L, Fini M, Giardino R. The microbial infection of biomaterials: A challenge for clinicians and researchers. A short review. J Appl Biomater Biomech. 2005 Jan-Apr;3(1):1-10. PMID 20799234
- [Background] Kurtz SM, Lau EC, Son MS, Chang ET, Zimmerli W, Parvizi J. Are We Winning or Losing the Battle With Periprosthetic Joint Infection: Trends in Periprosthetic Joint Infection and Mortality Risk for the Medicare Population. J Arthroplasty. 2018 Oct;33(10):3238-3245. doi: 10.1016/j.arth.2018.05.042. Epub 2018 Jun 1. PMID 29914821
- [Background] Aujla RS, Esler CN. Total Knee Arthroplasty for Osteoarthritis in Patients Less Than Fifty-Five Years of Age: A Systematic Review. J Arthroplasty. 2017 Aug;32(8):2598-2603.e1. doi: 10.1016/j.arth.2017.02.069. Epub 2017 Mar 3. PMID 28456563
- [Derived] de Lachica JCV, Reyes SSS, Urena JAP, Fragoso MAR. Decrease in acute periprosthetic joint infections incidence with vancomycin-loaded calcium sulfate beads in patients with non-modifiable risk factors. A randomized clinical trial. J ISAKOS. 2022 Dec;7(6):201-205. doi: 10.1016/j.jisako.2022.08.002. Epub 2022 Aug 13. PMID 35973626

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Inclusion critera for patients to complete enrolled protocol were: patients over 60 years old, no history of cephalosporine allergy, to have any of the non-modifiable risk factors, patients who accept blood transfusion. Patientes who are institutional entitled.
Groups:
- Calcium Sulfate Study Group: Group of members that will be submitted to prophylaxis with medicated calcium sulfate beads for hip or knee joint replacement
  Antibiotic local prophylaxis with medicated calcium sulfate beads: Antibiotic prophylaxis in patients with non-modifiable risk factors for periprosthetic joint infection. 3g of vancomycin mixed with Stimulan Kit (Biocomposites Ltd, United Kingdom) which includes 10 cc (20 g) of calcium sulfate hemihydrate powder
- Control Group: Group of members that will be submitted to classic prophylaxis for hip or knee joint replacement
  Classical parenteral antibiotic prophylaxis: Antibiotic prophylaxis in patients with non-modifiable risk factors for periprosthetic joint infection. 750 mgs of Intra Venous Ceftriaxone 20 minutes before joint replacement surgery and every 8 hours for 24 hours
Period: Overall Study
Arm/Group | Calcium Sulfate Study Group | Control Group
Started | 44 | 43
Completed | 43 | 40
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Sulfate Group | Control Group | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (8.14) | 77.3 (8.9) | 76.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 21 | 18 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 43 | 40 | 83
non-modifiable risk factors [Count of Participants; unit: Participants]
  Body Mass Index | 10 | 6 | 16
  Wound Drain, dehiscence or surgical active infecti | 2 | 4 | 6
  History of nosocomial infection | 3 | 3 | 6
  Prolonged surgical time | 3 | 4 | 7
  Decompensated Type 2 Diabetes Mellitus | 8 | 7 | 15
  Serum Albumin | 1 | 4 | 5
  Rheumatoid Arthritis | 2 | 5 | 7
  Blood transfusion Transoperative Bleeding | 7 | 5 | 12
  History of prosthetic surgery | 3 | 1 | 4
  Immunosuppression | 0 | 1 | 1
  Malignancy | 3 | 0 | 3
  Corticosteroid Therapy | 1 | 0 | 1
Location of Joint Prosthesis [Count of Participants; unit: Participants]
  KNEE | 17 | 21 | 38
  HIP | 26 | 19 | 45
Periprosthetic Joint Infection [Count of Participants; unit: Participants]
  With periprosthetic infection | 4 | 27 | 31
  Without periprosthetic infection | 39 | 13 | 52

OUTCOME MEASURES:

1. Primary Outcome: Partipants Achieving a Lower Hip or Knee Periprosthetic Joint Infection Rate With Local Versus Conventional Intravenous Antibiotic Prophilaxys, Measured With CRP, ERS in Serum and Sinovial Fluid Leukocytes , Over the 12-week Observation Period.
Description: Acute periprosthetic knee or hip infection was determined using CRP and ESR serum biomarkers, which are the most commonly published serum biomarkers in periprosthetic joint infection literature. The cut off point for CRP was considered 93mg/L and 44mm/hr for ESR. The serum biomarker sample was taken and evaluated on day 5 and weeks 4, 8 and 12. Leukocytes in synovial fluid are among the criteria for definition of periprosthetic joint infection with a cut off point above 12,800 cells/µL and were only included if serum biomarkers were elevated.
Time Frame: Day 5, Weeks 4, 8, and 12
Population: Patients who agreed to join the study and who met the selection criteria. After 3 moths presents or not periprosthetic joint infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Calcium Sulfate Group
Number analyzed (Participants) | 40 | 43
Participants
  With Periprosthetic Joint infection | 27 | 4
  Without periprosthetic infection | 13 | 39
Statistical Analysis 1: Comparison: Control Group vs Calcium Sulfate Group; H0.- There is no significant difference in the incidence of periprosthetic infection in patients with non-modifiable risk factors and prophylactic application of antibiotic loaded calcium sulfate compared with patients without prophylactic treatment with calcium sulfate. The presence of periprosthetic infection in both groups was evaluated by chi2 and Lambda tests for dichotomous nominal and qualitative variables with longitudinal direction and relative risk factor test; Test type: Superiority; p < 0.05, Chi-squared, Corrected; Risk Ratio (RR) = .049, 95% CI 2-sided [0.015 to 0.168] — For the Relative risk the control Study group was the numerator and control group denominator. In the 2X2 contingency table the rows correspond to groups and columns for the presence or abscence of periprosthetic infection

2. Secondary Outcome: Length of Stay as an Indicator of the Hospital Economic Burden
Description: The length of stay is an important indicator of efficiency and hospital economic burden. The reduction in number of hospitalization days results in lower risk of infection and less medication side effects and decreased need of hospital supplies. The difference in the average days of hospitalization between both groups indirectly represents the economic cost spent by the hospital.
Time Frame: Surgical procedure day to hospital discharge.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control Group | Calcium Sulfate Study Group
Number analyzed (Participants) | 40 | 43
Days | 15.25 (10.06) | 4.6 (4.62)
Statistical Analysis 1: Comparison: Control Group vs Calcium Sulfate Study Group; Lenght of stay was the variable that compares both groups and was a continous variable (t-test); Test type: Superiority; p < 0.01, t-test, 2 sided — The statistical test of t was performed for the variable length of hospital stay, finding a significant difference with a p value < 0.01

ADVERSE EVENTS:
Time Frame: 3 months after surgical procedure.
Description: Adverse mortality events from all causes, serious or other (non-serious) adverse events were monitored but none observed in the 3 months after the surgical procedure.
Arm/Group | Calcium Sulfate Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT03976466/Prot_SAP_ICF_001.pdf